CLINICAL TRIAL: NCT03914937
Title: Virtual Reality in Plastic Surgery: Pain Control and Augmented Satisfaction
Status: Completed | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1903-09
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Virtual Reality: Patients will wear a virtual reality device in addition to standard lidocaine/novocaine numbing agent
  Interventions: Other: Virtual reality
- Control Group: Music: Patients will listen to music in addition to standard lidocaine/novocaine numbing agent
  Interventions: Other: Music

INTERVENTIONS:
Other: Virtual reality — A virtual reality device will be worn over the eyes that allows the patient to feel that they are at a quiet seaside beach.
  Groups: Intervention Group: Virtual Reality
Other: Music — Music of the patient's choice will be played
  Groups: Control Group: Music

SUMMARY:
The study is looking at whether wearing a virtual reality device will help reduce pain and anxiety during minor procedures

DETAILED DESCRIPTION:
Patients who are undergoing minor plastic surgery procedures will be assigned to either wear a virtual reality device or to listen to music of their choice. Patients will still get the standard lidocaine/novocaine numbing agent. Patients will be asked questions about their anxiety level and pain level. Heart rate and blood pressure will be monitored as measures of anxiety and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for minor elective plastic surgery procedure
* Patients without cognitive, visual or hearing impairments

Exclusion Criteria:

* Patients with conditions that may prohibit participation or evaluation of the procedure (such as developmental delay)
* Lesions that involve portions of the head or face that will prohibit the use of VR goggles
* Severe vertigo
* Patients with nausea, vomiting, dementia, motion sickness, stroke, seizure and epilepsy and those placed in isolation (MRSA, VRE) were excluded.
* Patients who are pregnant
* Hearing or visually impaired
* Patients <18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for minor elective plastic surgery procedure
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Subjective Pain | 1 hour
  Subjective pain measured using the 11-point Numeric Rating Scale (NRS), which is widely employed and is a validated measure of pain (17) at the half way point and 1 minute after the procedure.The scale name is Pain Numeric Rating Scale (NRS) it is a validated scale for graphically measuring pain. The scale range is 0-10 (11 point scale). 0 is no pain. 10 is intolerable pain. The values on this scale will be averaged for each cohort.
Blood pressure | 1 hour
  Systolic and diastolic blood pressures (mmHg) at the half way point of the procedure as well as 1 minute after completion of the procedure. Blood pressure will be measured as a surrogate measure for objective pain. Blood pressures will be averaged for each cohort. The data will be collected by Dynamap automated Blood pressure monitor.
Heart rate | 1 hour
  Heart rate at the half way point of the procedure as well as 1 minute after completion of the procedure will be measured in beats per minute using pulse oximetry. Heart rate will be measured as a surrogate measure for objective pain. Heart rates will be averaged for each cohort.

SECONDARY OUTCOMES:
Anxiety | 1 hour
  Anxiety using an 11-point Numeric Rating Scale (NRS) at the half way point and 1 minute after completion of the procedure.The scale name for subjective anxiety measurement will be the Numeric Rating Scale (NRS) it is a validated scale for graphically measuring anxiety. The scale range is 0-10 (11 point scale). 0 is no pain. 10 is intolerable pain. The values on this scale will be averaged for each cohort.
Patient Satisfaction | 1 hour
  Patient satisfaction determined by the Global Rating Scale measured as 1-5 with 1 being unsatisfied and 5 being extremely satisfied. The Global Rating Scale (GRS) for patient satisfaction is a validated scale. These values will be averaged in each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Karim W Sadik, MD, Principal Investigator — The Guthrie Clinic; Crystal D Sadik, MD, Principal Investigator — The Guthrie Clinic; Nicholas Evertson, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sadik, K. , Miller, M. , Evertsen, N. , Sadik, C. and Bonatti, H. (2023) Virtual Reality in Surgery: Double Blind, Randomized Clinical Trial of Pain Control and Augmented Satisfaction. Surgical Science, 14, 456-467. doi: 10.4236/ss.2023.146050.
- See also: Link to publication doi: 10.4236/ss.2023.146050. — https://www.scirp.org/pdf/ss_2023063014591011.pdf